CLINICAL TRIAL: NCT01694680
Title: Intervention Study to Assess the Effect of Daily Consumption of a Lutein-enriched-egg Beverage on Maintenance of Visual Function in Subjects With Early Signs of Age-related Macular Degeneration
Brief Title: Intervention Trial in Early Age-related Macular Degeneration
Acronym: I-TEAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Newtricious R&D BV (Industry)
Collaborators: Sprim Advanced Life Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NWT-02/Human 4
Record Dates: First submitted 2012-09-25; First posted 2012-09-27 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Age-related Macular Degeneration (AMD)
Keywords: AMD; Lutein; Visual function; Early signs of AMD; AREDS-category 2
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lutein-enriched-egg beverage (Active Comparator): Powder in sachets is provided and dissolved to prepare Lutein-enriched-egg beverage
  Interventions: Dietary Supplement: Lutein-enriched-egg beverage (NWT-02)
- Placebo (Placebo Comparator): Powder in sachet to prepare beverage
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lutein-enriched-egg beverage (NWT-02) — Lutein, zeaxanthin and DHA-enriched-egg yolk combined with buttermilk beverage
  Arms: Lutein-enriched-egg beverage
Dietary Supplement: Placebo — color-, taste- and energy-matched powder without enriched egg-yolk
  Arms: Placebo

SUMMARY:
The purpose of the I-TEAM project is to assess whether there is a change in visual function and status of the retina after a year of intervention in subjects with early signs of Age-related Macular Degeneration.

ELIGIBILITY:
Inclusion Criteria:

* Early AMD (AREDS category 2)

  * many small drusen, or
  * a few intermediate-sized (63-124 micrometres in diameter) drusen, or
  * macular pigmentary changes

OR

* Intermediate AMD (AREDS category 3)

  * extensive intermediate sized (63-124 micrometres in diameter) drusen, or
  * at least one large (>125 micrometers in diameter) drusen or
  * geographic atrophy not involving the foveal centre
* men and women age ≥50 years
* BMI 18-35 kg/m2
* Vision ≥ 20/40 for Snellen visual acuity
* lutein intake of < 2 mg/day (including supplements)
* DHA intake of < 150 mg/day (including supplements)
* must be able to give written informed consent
* have normal hematologic parameters
* normal values of plasma albumin
* normal values for liver and kidney function
* no use of carotenoid, fish oil, or n3 fatty acid supplements (within 1 month of study start)

Exclusion Criteria:

* ocular media opacity (severe cataract)
* history of active small bowel disease or resection
* atrophic gastritis
* history of hyperlipidemia or screening values as follows (LDL > 5.33mmol/L or 205mg/dL; triglycerides > 4.52mmol/L or >400 mg/dL)
* hypertension (>150/90 mm Hg)
* diabetes mellitus (if also accompanied by signs of diabetic retinopathy)
* alcohol intake of >2 drinks/day or 14 drinks/week
* pancreatic disease
* dementia or Alzheimer's disease
* anemia, and bleeding disorders
* known allergy to egg or egg products
* known allergy to milk or milk products
* known allergy to cocoa or chocolate products
* known allergy to fish or fish oils
* lactose intolerance
* pregnancy or lactation
* diseases that interfere with fat absorption, e.g. colitis, celiac disease, Crohn's disease, cystic fibrosis (as determined by screening interview)
* medication or supplements that contain a significant level of carotenoids, including an amount of lutein of more than 0.25 mg per day within 1 month of the study start
* medications that interfere with fat absorption, e.g. bile sequestrants (as determined by screening interview)
* use of antipsychotic, anti manic, or dementia medications
* smoking or use of nicotine patches or gum (within the past 6 months)
* subjects having extremely high dietary intakes of carotenoids
* stroke, head injury with loss of consciousness or seizures
* for US and UK center: Non English speaking

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Visual function | 12 months

SECONDARY OUTCOMES:
Carotenoid levels | 12 months
  Levels of lutein and Zeaxanthin

CONTACTS AND LOCATIONS:
Overall Officials: E J Johnson, PhD, Principal Investigator — Jean Mayer USDA Human Nutrition Research Center on Aging (HNRCA), Boston
Locations (4):
- TUFTS University, Boston, Massachusetts, United States
- Universitäts Augenklinik - Bonn, Bonn, Germany
- Radboud University Hospital, Nijmegen, Netherlands
- Manchester Royal Eye Hospital - Manchester, Manchester, United Kingdom

REFERENCES:
- [Derived] Evans JR, Lawrenson JG. Antioxidant vitamin and mineral supplements for slowing the progression of age-related macular degeneration. Cochrane Database Syst Rev. 2023 Sep 13;9(9):CD000254. doi: 10.1002/14651858.CD000254.pub5. PMID 37702300